CLINICAL TRIAL: NCT02942563
Title: A Phase II Study of Total Neoadjuvant Therapy for Locally Advanced Rectal Cancer
Brief Title: Total Neoadjuvant Therapy for Locally Advanced Rectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016CRC R-001
Record Dates: First submitted 2016-10-21; First posted 2016-10-24 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Rectal Cancer
Keywords: Local Advanced Rectal Cancer; Total Neoadjuvant Therapy; FOLFOXIRI
MeSH Terms: conditions — Rectal Neoplasms | interventions — FOLFOXIRI protocol; Irinotecan; Oxaliplatin; Fluorouracil; Capecitabine

ARMS (1):
- FOLFOXIRI (Experimental): irinotecan* 165 mg/m² + oxaliplatin 85 mg/m² + leucovorin 200 mg/m² + 5-FU 2800 mg/m² cont. inf. 46h all on day 1 of each 2 weeks cycle
  Interventions: Drug: FOLFOXIRI

INTERVENTIONS:
Drug: FOLFOXIRI — Irinotecan* 165 mg/m² + oxaliplatin 85 mg/m² + leucovorin 200 mg/m² + 5-FU 2800 mg/m² cont. inf. 46h all on day 1 of each 2 weeks cycle for 4-6 cycles,
  Chemoradiation for patients who are not suitable to surgery:
  Pelvic radiotherapy(45Grey/25Fraction and 5.4Grey/3Fraction boost to the tumor bed) combined with capecitabine(625mg/m², bid po, d1-5, qw), and additional four cycles of modified FOLFOX6 (mFOLFOX6) or Oxaliplatin 135mg/m²plus Capecitabine 1.0/m² bid po(XELOX) of each 3 weeks cycle for 2 cycles chemotherapy before TME.
  All patients will receive 6-8 cycles of mFOLFOX6 or 4-5 cycles XELOX as adjuvant chemotherapy after TME.
  Other Names: Irinotecan; Oxaliplatin; 5-FU; Capecitabine

SUMMARY:
The concurrent neoadjuvant chemoradiation therapy is standard care for local advanced rectal cancer (LARC), however, this regimen may induce sorts of adverse events, and part of them even more severer. A number of pilot studies had shown high rate of complete resection after neoadjuvant chemotherapy alone, but the results did not increase the ratio of pathological complete response (pCR), which was associated with overall survival (OS). Here, the investigators adopt the three active cytotoxic agents (Fluorouracil, Oxaliplatin, Irinotecan, FOLFOXIRI) as the neoadjuvant chemotherapy regimen to replace the concurrent chemoradiation and to improve the ratio of pCR further.

DETAILED DESCRIPTION:
This is a multicenter, phase II trial to assess the efficacy/safety of triplet regimen (FOLFOXIRI) for patients with LARC. After 4 cycles of FOLFOXIRI and 2 weeks later, the patients will be evaluated by senior radiologist, oncologist and surgeon through pelvic MRI, CT and Positron Emission Computed Tomography (PET-CT). The patients will go to surgery (TME) if the tumor response is good enough to have complete resection under the decision of MDT,otherwise, the patients will receive pelvic radiotherapy(45Grey/25Fraction and 5.4Grey/3Fraction boost to the tumor bed) combined with capecitabine(625mg/M^2, bid po, d1-5, qw), and additional four cycles of modified FOLFOX6 (mFOLFOX6) or Oxaliplatin 135mg/m²plus Capecitabine 1.0/m² bid po(XELOX) of each 3 weeks cycle for 2 cycles chemotherapy before TME. All patients will receive 6-8 cycles of mFOLFOX6 or 4-5 cycles XELOX as adjuvant chemotherapy after TME.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 to 75 years at diagnosis
* Diagnosis of rectal adenocarcinoma
* ECOG status: 0～1
* Clinical stage II (T3-4, N0) or stage III (T1-4, N1-2)
* Adequate bone marrow, hepatic and renal function as assessed by the following laboratory requirements conducted within 7 days of starting study treatment:
* Leukocytes ≥ 4.0 x109/ L,
* Absolute neutrophil count (ANC) ≥ 2.0 x109/ L
* Platelet count ≥ 100 x109/ L,
* Hemoglobin (Hb) ≥ 9g/ dL.
* Total bilirubin ≤1.5 x the upper limit of normal (ULN).
* Alanine aminotransferase (ALT) ≤ 3 x ULN
* Aspartate aminotransferase (AST) ≤ 3 x ULN.
* Serum creatinine ≤ 1.5 x the ULN.
* Signed informed consent;

Exclusion Criteria:

* Patient had received pelvic radiotherapy
* Patient had received systemic chemotherapy
* Pregnant and Nursing women
* Had metastatic disease
* Uncontrolled co-morbid illnesses or other concurrent disease
* Patient had second malignant disease within 5 years
* Patients refused to signed informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Pelvic complete resection rate | Up to 10 weeks
  Pathologic confirmation

SECONDARY OUTCOMES:
The rate of local control | 3 years
  Imaging diagnosis
Disease free survival (DFS) | 3 years
  Imaging diagnosis
Overall survival | 3 years
  Record document
The rate of receive chemoradiation | Up to 10 weeks
  Record document
The rate of clinical complete response after 4 cycles of FOLFOXIRI | Up to 10 weeks
  Imaging diagnosis
The rate of pathological complete response after 4 cycles of FOLFOXIRI | Up to 10 weeks
  Pathologic confirmation
The incidence of >=3 grade adverse events | 2 years
  Common Terminology Criteria for Adverse Events v3.0 (CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Ming Ye, Master, Principal Investigator — Locations: China, Shanghai Shanghai Jiaotong University School of Medicine, Renji Hospital
Locations (1):
- Ethics Committee of Renji Hospital, School of Medicine,Shanghai Jiaotong University, Shanghai, Shanghai Municipality, China